CLINICAL TRIAL: NCT01346982
Title: Drug Interactions Between Silimarine And Darunavir/Ritonavir
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundación FLS de Lucha Contra el Sida, las Enfermedades Infecciosas y la Promoción de la Salud y la Ciencia (Other)
Collaborators: IrsiCaixa (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SILIDAR; 2010-021159-25
Record Dates: First submitted 2011-04-18; First posted 2011-05-04 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2011-09

CONDITIONS: HIV
Keywords: Darunavir; Silimarine; interaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Silimarine (Experimental): darunavir + ritonavir + silimarine
  Interventions: Drug: Silimarine

INTERVENTIONS:
Drug: Silimarine — darunavir/ritonavir 600/100 mg + silimarine (150 mg every 8 hours)

SUMMARY:
This is a clinical trial to characterize drug interactions between silimarine and the protease inhibitor darunavir/ritonavir.

DETAILED DESCRIPTION:
The silimarine is the main component of milk thistle (Sylibum marianum), a medicinal herb which, due to its attributed hepatoprotective properties, is widely used by HIV infected patients

15 patients on stable antiretroviral therapy including darunavir/ritonavir 600/100 mg twice a day during four weeks will be enrolled. After their inclusion in the study, patients will receive treatment with silimarine (150 mg every 8 hours) from day 1 until two weeks later (day 14). On days 0 and 14, blood samples will be drawn immediately before and 1, 2, 4, 6, 8, 10 and 12 hours after the administration of darunavir/ritonavir, and darunavir and ritonavir concentrations in plasma will be determined by high performance liquid chromatography using a validated method.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving antiretroviral therapy containing darunavir / ritonavir at the approved dose of 600/100 mg twice daily for at least 4 weeks
* HIV viral load in plasma <50 copies / mL
* Absence of acute infections and / or tumors in the three months prior to inclusion.
* Subject able to follow the treatment period, without suspicion of poor adherence in previous antiretroviral treatments.

Exclusion Criteria:

* Any clinical or historical observation that could interfere with the pharmacokinetics of medications, such as gastrointestinal illness or surgery (except for herniotomy and appendectomy), changes in the composition of plasma proteins, some indication of hepatic or renal dysfunction.
* Active alcohol consumption (> 50 g / day) or illicit drugs (except cannabis).

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2011-03; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve during the dosing interval (AUC0-12) of darunavir | DAY 0, day 14

SECONDARY OUTCOMES:
Area under the plasma concentration-time curve during the dosing interval (AUC0-12) of ritonavir | DAY 0, day 14
Darunavir and ritonavir clearance (CL/F) | DAY 0, day 14
  Change from day 0 in Darunavir and ritonavir clearance at day 14
Darunavir and ritonavir volume of distribution (V/F) | DAY 0, day 14
  Change from day 0 in Darunavir and ritonavir volume of distribution at day 14
Darunavir and ritonavir elimination half-life (t1/2) of darunavir and ritonavir | DAY 0, day 14
Darunavir and ritonavir trough concentration in plasma | DAY 0, day 14
Adverse events and laboratory abnormalities | DAY 0, 14, 28
  Number of patients with adverse events and laboratory abnormalities grade 3 or 4

CONTACTS AND LOCATIONS:
Locations (1):
- Lluita contra la Sida Foundation, HIV Unit, Badalona, Barcelona, Spain